CLINICAL TRIAL: NCT03591276
Title: A Phase 1b Study of Combination Chemo-immunotherapy With Pegylated Liposomal Doxorubicin (Doxil/Caelyx) and Pembrolizumab (Keytruda) in Metastatic Endocrine-resistant Breast Cancer
Brief Title: Phase 1b Study of Pegylated Liposomal Doxorubicin and Pembrolizumab in Endocrine-resistant Breast Cancer
Acronym: KEYDOX
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 310-17-SZMC
Record Dates: First submitted 2018-06-26; First posted 2018-07-19 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; immune check point inhibitors; chemotherapy; liposomal doxorubicin; pharmacokinetics; Anti-PD1 antibodies
MeSH Terms: conditions — Breast Neoplasms | interventions — Antineoplastic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab and PLD (Experimental): Cohort S1: IV pembrolizumab 200 mg flat dose with IV PLD 30 mg/m2 every 3 weeks.
  Reduced Dose Cohort (R1)*: IV pembrolizumab 200 mg flat dose with IV PLD 24 mg/m2 every 3 weeks.
  *Subjects will be recruited into the R1 cohort only if DLT is reported in 2 or more subjects during the first 2 cycles of treatment in the first 6 patients of the S1 cohort.
  Interventions: Drug: Chemotherapy Drugs, Cancer

INTERVENTIONS:
Drug: Chemotherapy Drugs, Cancer — IV pembrolizumab 200 mg flat dose with IV PLD 30 mg/m2 (chemotherapy drugs) every 3 weeks in eligible breast cancer patients.
  Other Names: Immunotherapy Antibodies, Cancer

SUMMARY:
Very few patients with endocrine-resistant, hormone-receptor positive metastatic breast cancer respond to single agent immunotherapy. Responses to chemotherapy are usually of short duration. Combining immunotherapy with chemotherapy that has minimal immunosuppressive effect, it may be possible to achieve higher response rates while keeping the immune-associated pattern of long durations of response.

This will be a single-center phase 1b study to evaluate the tumor response and appropriate dose of a chemo-immunotherapy regime consisting of treatment with pegylated liposomal doxorubicin (PLD) and pembrolizumab-based in endocrine-resistant breast cancer (ERBC) patients.

Up to 15 female patients, ages 18 and above, with pathological diagnosis of breast cancer, estrogen receptor (ER) positive, human epidermal growth factor receptor 2 (HER2-) negative subtype, stage III non-operable, or stage IV disease, who have received at least two lines of hormonal therapy, one of which included aromatase inhibitors will be eligible for enrollment to this single arm study.

DETAILED DESCRIPTION:
This will be a single-center phase 1b study to evaluate the tumor response and appropriate dose of combined treatment with pembrolizumab and pegylated liposomal doxorubicin (PLD) in endocrine-resistant breast cancer (ERBC) patients.

Female patients, ages 18 and above, with pathological diagnosis of breast cancer, estrogen receptor (ER) positive, human epidermal growth factor receptor 2 (HER2-) negative subtype, stage III non-operable, or stage IV disease, who have received at least two lines of hormonal therapy, one of which included aromatase inhibitors will be eligible for enrollment to the study.

The total number of patients in the study will be 15 patients. The study diagram is shown in Figure 1. After signing the informed consent, eligible subjects will be successively assigned, in order of accrual, to a dosing cohort. Six subjects will be enrolled in the Start Cohort (Cohort S1), and receive: intravenous (IV) pembrolizumab 200 mg flat dose with IV pegylated liposomal doxorubicin (PLD) 30 mg/m2, every 3 weeks. Toxicity will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events Ver. 4.0 (NCI-CTCAE).

If during the first 2 cycles of treatment (the first 6 weeks) in the Start Cohort (Cohort S1), up to one subject out of the 6 in the cohort will develop a dose-limiting toxicity (DLT; defined as grade-4 hematological adverse events (AEs), or grade 3 non-hematological AEs [stomatitis, hand and foot syndrome] in the first 2 cycles), the drug combination's safety profile will be deemed acceptable and up to 9 more subjects will be recruited in the cohort (Expanded Start Cohort S1) and will receive the same dose to help establish the rate of Tumor Response and to confirm safety.

If during the first 2 cycles of treatment in the Start Cohort (Cohort S1) a DLT will be observed in 2 or more patients out of the initial 6 patients enrolled into this cohort, Cohort S1 will be discontinued, and a Reduced Dose Cohort (Cohort R1), will be accrued where the dose of PLD will be reduced by 20% to 24 mg/m2 (IV pembrolizumab 200 mg flat dose with IV PLD 24 mg/m2 every 3 weeks). Initially, 6 patients will be accrued to Cohort R1. If during the first 2 cycles of treatment (the first 6 weeks) in the Reduced Dose Cohort (Cohort R1), up to one subject out of the 6 in the cohort will develop a DLT, the drug combination's safety profile will be deemed acceptable and up to 7 more subjects will be recruited in the cohort (Expanded Reduced Cohort R1) to help establish the rate of Tumor Response and to confirm safety of the reduced dose.

If during the first 2 cycles of treatment in Cohort R1, a DLT would be again observed in 2 or more subjects, the study will be terminated (refer to Figure 1 for the study diagram).

Note: Only the first 2 cycles will be considered for safety clearance of any Cohort. If an additional DLT occurs in the 3rd cycle, the dose will be individually modified if the affected patient has stable disease (SD) or partial response/complete response (PR/CR), and the patient will continue to the extended phase of the study.

The 3 first cycles of treatment (first 9 weeks) constitute the main phase of the study during which most of the study objectives will be reached (safe dose clearance, tumor response rate characterization of DLT's, pharmacokinetic [PK] analysis of PLD). Patients will return to the study center on days 7 and 14 of cycles 1, 2 and 3, for monitoring assessments and for clinical laboratory evaluations. Blood samples will be collected on study visits for measurement of PLD concentrations at various time points during cycle 1. For each subject, subsequent dosing will take place 21 days after the previous treatment, provided patients are deemed fit to be dosed again.

For responding or stable patients, the extended phase of the study consists of 9 additional cycles (27 more weeks) during which further safety information, duration of response, progression-free survival (PFS) time, and other pertinent data will be collected. During both phases of the study and beyond, information on survival and post-study treatments will be collected until death. Information on potentially predictive biomarkers of treatment response (and duration of response) will be gathered all along the study.

All patients receiving two or more cycles will be followed-up for survival until death. Study treatment may continue until disease progression, unacceptable toxicity, patient refusal, patient loss to follow up, or termination of the study by the Sponsor or Investigator, whichever comes first. Pembrolizumab may be continued beyond disease progression. PLD will not be continued beyond disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Have pathological diagnosis of breast cancer, ER positive (%ER+ cells≥1%, Allred score ≥3), Her2 negative subtype, locally advanced (stage III non-operable), or metastatic (stage IV) disease.
2. Have measurable disease on computed tomography (CT) or positron emission tomography-computed tomography (PET-CT) scan.

2. Be 18 years of age on day of signing informed consent. 3. Have measurable disease based on RECIST 1.1. 4. Have Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1. 5. Have an estimated life expectancy of at least 3 months. 6. Demonstrate adequate organ function as defined in Table 1. All screening labs should be performed within 10 days of treatment initiation.

7. Have received at least two lines of hormonal therapy, one of which had included aromatase inhibitors.

8. May have received none or up to 2 lines of chemotherapy (excluding any chemotherapy given in adjuvant or pre-operative-neoadjuvant settings).

9. Have a ≥21-day treatment-free interval from chemotherapeutic treatment. 10. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

11. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2, for the course of the study through 120 days after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

12. Understanding of study procedures and willingness to comply throughout the entire course of the study and to provide written informed consent.

Exclusion Criteria:

1. Has known hypersensitivity to the study drugs or to any of their excipients.
2. Has congestive heart failure (New York Heart Association [NYHA] Class IV) or left ventricular ejection fraction (LVEF) ≤40%.
3. Has chronic obstructive pulmonary disease (COPD) >Stage 3 (forced expiratory volume in 1 second [FEV1] <50%, forced expiratory volume 1/forced vital capacity [FEV1/FVC] <70%).
4. Has cirrhosis (Child-Pugh Class C score).
5. Has serum albumin level < 2.5 g/dl.
6. Has a known history of HIV (HIV 1/2 antibodies).
7. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
8. Has evidence of active bleeding or bleeding diathesis.
9. Concomitant use of any other chemotherapy (except for PLD) or hormonal therapy during the study
10. Uncontrolled ascites (defined as 2 or more palliative taps within 30 days of screening).
11. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
12. Continuous steroid treatment for other than brain metastases requiring daily corticosteroid dose ≥ 10 mg prednisone or corticosteroid-equivalent per day.
13. Anthracycline treatment (doxorubicin, epirubicin, mitoxantrone, PLD) in metastatic setting.
14. Less than 6 months from last treatment with anthracyclines in adjuvant or neo-adjuvant setting.
15. Use of any investigational drug within 28 days prior to study entry.
16. Diagnosis of any other malignancy within 5 years prior to registration, except for adequately treated basal cell or squamous cell skin cancer, superficial melanoma, or carcinoma in situ of the breast or of the cervix.
17. Severe gastrointestinal conditions such as clinical or radiological evidence of bowel obstruction within 4 weeks prior to study entry, or uncontrolled diarrhea in the last 4 weeks prior to enrollment.
18. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
19. Has a diagnosis of immunodeficiency or is receiving any immunosuppressive therapy (except for prednisone ≤10 mg/day or equivalent) within 7 days prior to the first dose of trial treatment.
20. Has a known history of active Bacillus Tuberculosis.
21. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to agents administered more than 4 weeks earlier.
22. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 3 weeks prior to study Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to a previously administered agent.

    Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

    Note: If the subject underwent major surgery, she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
23. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin or melanoma that have undergone potentially curative therapy or in situ cervical or bladder cancer.
24. Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases are eligible for recruitment provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and may be receiving dexamethasone at a dose ≤4 mg/day prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
25. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
26. Has a known history of, or any evidence of active, non-infectious pneumonitis.
27. Has an active serious infection or an active infection requiring systemic therapy.
28. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
29. Has a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
30. Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
31. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
To establish a safe dose of PLD when delivered in combination with pembrolizumab | At the end of Cycle 2 (day 42), each cyle is 21 days
  A dose will be considered safe when the number of Participants With Treatment-Related Adverse Events grades 3 or 4, as assessed by CTCAE v4.0, will be less than 2 per 6-patient cohort. Our hypothesis is that treatment with pembrolizumab will be compatible with the standard recommended dose of PLD,
To evaluate the Tumor Response Rate according to Response Evaluation Criteria in Solid Tumors (RECIST) after 9 weeks (3 cycles) of treatment in patients with measurable disease. | At the end of Cycle 3 (day 63), each cycle is 21 days
  Th response rate will be evaluated after 9 weeks (3 cycles) by RECIST. Our hypothesis is that the response rate of the combination will be higher than expected from each agent alone.

SECONDARY OUTCOMES:
To evaluate the safety and DLT of the PLD and pembrolizumab combination, as indicated by the number of study participants with treatment-related Adverse Events, and the class of Adverse Events as assessed by CTCAE v4.0. | At the end of Cycle 2 (day 42), each cycle is 21 days
  The safety profile of PLD and pembrolizumab will be evaluated by the number of study participants with treatment-related Adverse Events, and the class of Adverse Events as assessed by CTCAE v4.0. Our hypothesis is that it will remain unchanged when given in combination, as compared to what expected for each drug alone.
To characterize the PK of PLD when delivered in combination with pembrolizumab, by measuring and comparing the Area under the curve (AUC) for doxorubicin (liposomal) obtained during Cycles 1 and 3. | During Cycle 1 (between days 1 and 22), and Cycle 3 (between days 42 and 63), each cycle is 21 days
  The PK of PLD will be evaluated by quantitation of doxorubicin (liposomal) in plasma samples and calculation of the AUC. Hypothesis: The PK profile of PLD may be modified by pembrolizumab during the course of therapy due to indirect effects on the mononuclear-phagocyte system (MPS) which plays an important role in PLD clearance. This will translate into a decrease or increase of AUC when the results of the 1st and 3rd cycles are compared.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto A Gabizon, MD, PhD, Principal Investigator — Shaare Zedek MC
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] O'Brien ME, Wigler N, Inbar M, Rosso R, Grischke E, Santoro A, Catane R, Kieback DG, Tomczak P, Ackland SP, Orlandi F, Mellars L, Alland L, Tendler C; CAELYX Breast Cancer Study Group. Reduced cardiotoxicity and comparable efficacy in a phase III trial of pegylated liposomal doxorubicin HCl (CAELYX/Doxil) versus conventional doxorubicin for first-line treatment of metastatic breast cancer. Ann Oncol. 2004 Mar;15(3):440-9. doi: 10.1093/annonc/mdh097. PMID 14998846
- [Result] Tahover E, Patil YP, Gabizon AA. Emerging delivery systems to reduce doxorubicin cardiotoxicity and improve therapeutic index: focus on liposomes. Anticancer Drugs. 2015 Mar;26(3):241-58. doi: 10.1097/CAD.0000000000000182. PMID 25415656
- [Result] Rios-Doria J, Durham N, Wetzel L, Rothstein R, Chesebrough J, Holoweckyj N, Zhao W, Leow CC, Hollingsworth R. Doxil synergizes with cancer immunotherapies to enhance antitumor responses in syngeneic mouse models. Neoplasia. 2015 Aug;17(8):661-70. doi: 10.1016/j.neo.2015.08.004. PMID 26408258
- [Result] Gabizon AA, Patil Y, La-Beck NM. New insights and evolving role of pegylated liposomal doxorubicin in cancer therapy. Drug Resist Updat. 2016 Nov;29:90-106. doi: 10.1016/j.drup.2016.10.003. Epub 2016 Oct 29. PMID 27912846